CLINICAL TRIAL: NCT00027794
Title: Radical Prostatectomy for Locally Advanced Prostate Cancer. A Feasibility Study
Brief Title: Radical Prostatectomy in Treating Patients With Locally Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-30001; EORTC-30001
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Procedure: conventional surgery

SUMMARY:
RATIONALE: Radical prostatectomy may be an effective treatment for locally advanced prostate cancer.

PURPOSE: Phase II trial to study the effectiveness of radical prostatectomy in treating patients who have locally advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the success rate of radical prostatectomy in patients with locally advanced adenocarcinoma of the prostate.
* Determine the serious toxic event rate of this surgery in these patients.
* Determine the pN status of patients treated with this surgery.
* Determine the percentage of patients found to have organ-confined tumors (pT2) after undergoing this surgery.
* Determine the 2-year prostate-specific antigen-free survival rate of patients treated with this surgery.
* Determine the surgical morbidity rates of patients treated with this surgery.

OUTLINE: This is a multicenter study.

Patients undergo limited pelvic lymphadenectomy and then radical retropubic prostatectomy.

Patients who are found to have pN-positive disease receive further treatment according to the investigator's discretion. Patients with pN0 disease are followed every 3 months for 1 year and then every 4 months for 1 year.

PROJECTED ACCRUAL: A total of 32-74 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Unilateral cT3a, cN0, M0
* Well or moderately differentiated tumor

  * Gleason score no greater than 7 (4 plus 3 or 3 plus 4)
* Total serum prostate-specific antigen no greater than 20 ng/mL (Hybritech equivalent)

PATIENT CHARACTERISTICS:

Age:

* 70 and under

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 9 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times normal
* ALT or AST less than 3 times normal
* PT and PTT normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No preexisting uncontrolled cardiac disease, signs of cardiac failure, or rhythm disturbances requiring therapy
* No myocardial infarction within the past 6 months

Pulmonary:

* No gross abnormalities on chest x-ray

Other:

* No other disease that would preclude surgery
* No other prior malignancy except adequately treated basal cell skin cancer
* No other concurrent primary malignancy
* No psychological, familial, sociological, or geographical condition that would preclude compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No prior hormonal therapy that would affect assessment of clinical T staging, margin positivity, or definitive pT staging

Radiotherapy:

* No prior pelvic radiotherapy that would affect surgical resectability and perioperative morbidity

Surgery:

* No prior surgery in the small pelvis (vascular surgery, mesh graft hernia repair, any surgery for benign prostatic hypertrophy, or transurethral resection of prostate) that would preclude prostatectomy

Max Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-09; Primary Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hein van Poppel, MD, PhD, Study Chair — University Hospital, Gasthuisberg
Locations (5):
- Belgium (2):
  - Virga Jesse Hospital, Hasselt
  - U.Z. Gasthuisberg, Leuven
- Italy (2):
  - Istituto Scientifico H. San Raffaele, Milan
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Martin Faculty Hospital, Martin, Slovakia

REFERENCES:
- [Result] Van Poppel H, Vekemans K, Da Pozzo L, Bono A, Kliment J, Montironi R, Debois M, Collette L. Radical prostatectomy for locally advanced prostate cancer: results of a feasibility study (EORTC 30001). Eur J Cancer. 2006 May;42(8):1062-7. doi: 10.1016/j.ejca.2005.11.030. Epub 2006 Apr 18. PMID 16624554